CLINICAL TRIAL: NCT00172484
Title: North Taiwan Stroke Center for Prevention and Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 9361700808
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Cerebrovascular Accident
Keywords: cerebrovascular accident; stroke center; stroke team; intensive care of stroke; rehabilitation of stroke
MeSH Terms: conditions — Stroke | interventions — Early Intervention, Educational; Nursing Evaluation Research; Rehabilitation

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Procedure: education program — A well-designed questionnaire concerning about awareness of stroke symptoms, knowledge, and management was done in adults of stroke victims' family members and general population.
Procedure: nursing program — To establish a systemic stroke prevention, education protocol
Procedure: rehabilitation program — From a sample of 648 stroke patients who were referred to rehabilitation between November 2002 and October 2002, 345 charts were successfully reviewed. Besides, 126 subjects were randomly selected and successfully contacted for telephone follow-up; and data from 87 subjects of telephone survey were included for statistical analysis. Comparison of functional status between early rehabilitation and ordinary scheduled rehabilitation for acute stroke patients was done from admission to 3 months after stroke onset. The efficacy of early application of electric stimulation for the upper paralyzed extremity was performed.

SUMMARY:
The Northern Taiwan Stroke Center for Prevention and Treatment Project is a single medical center, 3-year, multipurpose study. The aims of this study are (1) to set up a multidisciplinary stroke team in a well-designed stroke center for stroke care; (2) to establish a systemic stroke prevention / education protocol based on people's awareness of stroke; and (3) to create a better stroke rehabilitation protocol and pathway.there are three components in rehabilitation projects. First, we want to identify potential factors related to functional outcome in patients with stroke before and after stroke center. Second, we want to compare the functional outcome in patients who admit to the stroke center as to those admitted to the general ward. Third, we want to investigate the effect of electrical stimulation on upper limb function in patient with acute stroke.

ELIGIBILITY:
Inclusion Criteria:

* acute stroke
* age > 18 y/o
* consult rehabilitation
* client or agent can sign a letter of consent

Exclusion Criteria(for rehabilitation protocol):

* contraindication of electrical stimulation(pacemaker implant, severe arrhythmia, malignant cancer, wound on stimulation site)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2005-01; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Bureau Of Health Promotion,Department of Health , R.O.C. | 2003/08/29；2004/02/02；2004/08/26；2004/12/03；2005/06/12；2005/11/22

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Keung Yip, Study Chair — Department of Neurology, National Taiwan Univisity Hospital
Locations (1):
- Stroke Intensive Care Unit, Taipei, Taiwan